CLINICAL TRIAL: NCT02407106
Title: Efficacy of Streptococcus Salivarius BLIS (Bacteriocin-like Inhibitory Substance) K12 as Preventive Measure for Rheumatic Children.
Brief Title: Efficacy of BLIS K12 as Preventive Measure for Rheumatic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Dr Yael Garty MD, MD, Kaplan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 027-15-KMC
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatic Fever
Keywords: BLIS K12; streptococcus
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BLIS K12 treatment (Experimental): Once daily tablet of Streptococcus Salivarius BLIS K 12 to be slowly dissolved orally every evening for six month
  Interventions: Dietary Supplement: Streptococcus Salivarius BLIS K12

INTERVENTIONS:
Dietary Supplement: Streptococcus Salivarius BLIS K12 — Once daily tablet of BLIS K 12 to be slowly dissolved orally every evening.
  Other Names: Bio-BLIS

SUMMARY:
The purpose of this study is to determine whether daily treatment with Streptococcus Salivarius BLIS K-12 prevents streptococcal throat infection in children that have had an episode of rheumatic fever.

DETAILED DESCRIPTION:
Children diagnosed with Rheumatic fever are currently given preventive streptococcal treatment with either monthly IM (intramuscular injection) Penicillin or daily oral Penicillin.

This preventive treatment is recommended for years until the child is 20 y old or even later. The compliance rate for this treatment declines significantly with time (the injections are painful) and even with good adherence the prevention is not complete.

In the last few years a new product licensed as "BLIS K-12" has been developed and approved by FDA as GRAS (generally recognized as safe) status from 2011.

This probiotic treatment prevents the pathogenic Strep A from adhering to the throat of the child thus preventing the infection. This kind of prevention is better for the long run for the patient and for the surrounding, It is better tolerated, is effective even if a dose is skipped or missed is not painful and is tasty to the children.

So the investigators assumption is that giving this product to children instead of Penicillin either orally or intramuscularlly will be better tolerated thus give a better protection profile with much less side effects.

The investigators will be giving BLIS K-12 to those children on the trial on a daily basis for 6 autumn-winter months instead of Penicillin and will monitor the children by monthly throat swabs. The investigators will also obtain Anti Streptolysin blood test at the end of the period from all participants to evaluate possible Strep encounters.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatic heart disease with recommended strep prophylaxis

Exclusion Criteria:

* less than one year from first diagnosis
* refusal to take the tablets

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
number of Strep throat infections while in study | six month

CONTACTS AND LOCATIONS:
Overall Officials: Yael Garty, MD, Principal Investigator — Attending physician

REFERENCES:
- [Background] May G, Wilson MG, Lubschez R. Recurrence rates in rheumatic fever. JAMA. 1944, Vol. 126, 8, pp. 477-480.
- [Background] Spagnuolo M, Pasternack B, Taranta A. Risk of rheumatic-fever recurrences after streptococcal infections. Prospective study of clinical and social factors. N Engl J Med. 1971 Sep 16;285(12):641-7. doi: 10.1056/NEJM197109162851201. No abstract available. PMID 4254612
- [Background] FEINSTEIN AR, WOOD HF, EPSTEIN JA, TARANTA A, SIMPSON R, TURSKY E. A controlled study of three methods of prophylaxis against streptococcal infection in a population of rheumatic children. II. Results of the first three years of the study, including methods for evaluating the maintenance of oral prophylaxis. N Engl J Med. 1959 Apr 2;260(14):697-702. doi: 10.1056/NEJM195904022601405. No abstract available. PMID 13644570
- [Background] Lue HC, Wu MH, Hsieh KH, Lin GJ, Hsieh RP, Chiou JF. Rheumatic fever recurrences: controlled study of 3-week versus 4-week benzathine penicillin prevention programs. J Pediatr. 1986 Feb;108(2):299-304. doi: 10.1016/s0022-3476(86)81009-5. PMID 3511209
- [Background] John D.F. Hale, John R. Tagg, and Philip A. Wescombe. BLIS-producing probiotics targeting the oral cavity. Microbiology Australia. 2012, Vol. 33, 3, pp. 103-105.
- [Background] Barretto C, Alvarez-Martin P, Foata F, Renault P, Berger B. Genome sequence of the lantibiotic bacteriocin producer Streptococcus salivarius strain K12. J Bacteriol. 2012 Nov;194(21):5959-60. doi: 10.1128/JB.01268-12. PMID 23045482
- [Background] J. Tagg, P. Wescombe , J. Burton. Oral streptococcal BLIS: Heterogeneity of the effector molecules and potential role in the prevention of streptococcal infections. International Congress Series. 2006, Vol. 128, pp. 347-350.
- [Background] Wescombe PA, Upton M, Dierksen KP, Ragland NL, Sivabalan S, Wirawan RE, Inglis MA, Moore CJ, Walker GV, Chilcott CN, Jenkinson HF, Tagg JR. Production of the lantibiotic salivaricin A and its variants by oral streptococci and use of a specific induction assay to detect their presence in human saliva. Appl Environ Microbiol. 2006 Feb;72(2):1459-66. doi: 10.1128/AEM.72.2.1459-1466.2006. PMID 16461700
- [Background] Di Pierro F, Colombo M, Zanvit A, Risso P, Rottoli AS. Use of Streptococcus salivarius K12 in the prevention of streptococcal and viral pharyngotonsillitis in children. Drug Healthc Patient Saf. 2014 Feb 13;6:15-20. doi: 10.2147/DHPS.S59665. eCollection 2014. PMID 24600248
- [Background] Burton JP, Chilcott CN, Wescombe PA, Tagg JR. Extended Safety Data for the Oral Cavity Probiotic Streptococcus salivarius K12. Probiotics Antimicrob Proteins. 2010 Oct;2(3):135-44. doi: 10.1007/s12602-010-9045-4. PMID 26781236
- [Background] Burton JP, Cowley S, Simon RR, McKinney J, Wescombe PA, Tagg JR. Evaluation of safety and human tolerance of the oral probiotic Streptococcus salivarius K12: a randomized, placebo-controlled, double-blind study. Food Chem Toxicol. 2011 Sep;49(9):2356-64. doi: 10.1016/j.fct.2011.06.038. Epub 2011 Jun 21. PMID 21722694
- [Background] Di Pierro F, Donato G, Fomia F, Adami T, Careddu D, Cassandro C, Albera R. Preliminary pediatric clinical evaluation of the oral probiotic Streptococcus salivarius K12 in preventing recurrent pharyngitis and/or tonsillitis caused by Streptococcus pyogenes and recurrent acute otitis media. Int J Gen Med. 2012;5:991-7. doi: 10.2147/IJGM.S38859. Epub 2012 Nov 30. PMID 23233809